CLINICAL TRIAL: NCT00984932
Title: The Effect of Rosuvastatin on Vascular Dysfunction and Inflammatory Markers in Systemic Sclerosis-related Pulmonary Hypertension: Randomized, Double-Blind Placebo-Controlled Trial
Brief Title: Effect of Rosuvastatin on Systemic Sclerosis-related Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Dr Anna Abou-Raya, Faculty of Medicine, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed116613963
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; pulmonary hypertension; rosuvastatin
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg of rosuvastatin daily
  Other Names: Statin, Crestor

SUMMARY:
Although the aetiology of SSc-PAH remains elusive, vascular dysfunction seems to be the initial event and statins through their vasculoprotective effect might be of value in the treatment armamentarium of PAH related to SSc.

The aim was to assess the efficacy of rosuvastatin in ameliorating vascular dysfunction and in the management of SSc-related PAH.

DETAILED DESCRIPTION:
Background: Pulmonary arterial hypertension (PAH) is an acknowledged devastating complication of systemic sclerosis (SSc); difficult to manage with a poor prognosis.

Although the aetiology of SSc-PAH remains elusive, vascular dysfunction seems to be the initial event.

Statins, through their pleotropic effects might be of value in the treatment armamentarium of PAH related to SSc.

Objectives: The aim was to assess the efficacy of rosuvastatin in ameliorating vascular dysfunction and in the management of SSc-related PAH.

Methods: Forty SSc patients fulfilling the ACR criteria for the classification of SSc diagnosis and having PAH were recruited.

All SSc patients underwent transthoracic echocardiography and the six minute walk test (SMWT).

Patients were randomized into 2 groups; the first group (n = 23) were assigned to receive 40mg of rosuvastatin and the second group (n = 23) received placebo for 6 months.

The levels of endothelial dysfunction and inflammatory markers were assayed at baseline and after 6 months of therapy. Outcome measures assessed included exercise capacity (SMWT), MPAP, WHO functional class change, tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) class III
* A mean pulmonary artery pressure (mPAP) of > 30mmHg at rest

Exclusion Criteria:

* Smoking
* Diabetes mellitus
* Hypercholesterolemia
* Hypertension
* Cardiac insufficiency
* Coexisting hepatic and renal diseases
* Use of drugs known to interact with statins.
* Patients with severe interstitial lung fibrosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
exercise capacity measured by the SMWT, mPAP and WHO functional class change | At baseline and After 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Alexandria Governorate, Egypt